CLINICAL TRIAL: NCT07142642
Title: A Phase 1, Randomized, Placebo-controlled, Double-blind, Single-dose Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Teprotumumab (AMG 632) Administered Intravenously in Healthy Chinese Participants
Brief Title: A Study to Evaluate Pharmacokinetics, Safety, and Tolerability of Teprotumumab (AMG 632) Administered Intravenously in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20240181
Record Dates: First submitted 2025-08-25; First posted 2025-08-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Healthy Chinese participants; Thyroid eye disease; TED; Thyroid-associated ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Teprotumumab (Experimental): Participants will be randomized 3:1 to receive a single IV infusion of teprotumumab or placebo on Day 1.
  Interventions: Drug: Teprotumumab
- Placebo (Placebo Comparator): Participants will be randomized 3:1 to receive a single IV infusion of teprotumumab or placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teprotumumab — Administered via IV infusion.
  Other Names: Tepezza; AMG 632
  Arms: Teprotumumab
Drug: Placebo — Administered via IV infusion.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of teprotumumab after a single intravenous (IV) infusion of teprotumumab in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent.
2. Participants must be a resident in mainland China, and of Chinese ancestry (participants whose parents within 3 generations are of Chinese ancestry).
3. Male or female participants, between 18 and 60 years of age (inclusive). Female participants must be of nonchildbearing potential.
4. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations.
5. Body mass index between 18 and 27 kg/m^2 (inclusive) and minimum weight of 55 kg .

Exclusion Criteria:

1. History or evidence of clinically significant disorder, condition, or disease.
2. History of diabetes. (regardless of type with the exception of history of gestational diabetes). Hemoglobin A1C greater than or equal to 6.5% (greater than or equal to 48 mmol/mol).
3. Fasting glucose level (after at least an 8-hour fast) > 126 mg/dL (> 7 mmol/L).
4. History of or ongoing hearing impairment.
5. History of any autoimmune disease, inflammatory bowel disease, or TED.
6. History or evidence of ECG-findings.
7. Systolic blood pressure ≥ 140 mmHg or < 90 mmHg, or diastolic blood pressure ≥ 90 mmHg or < 50 mmHg, or pulse > 100 bpm or < 50 bpm , at screening or check-in.
8. History of relevant drug and/or food allergies.
9. Poor peripheral venous access and/or unable to receive IV infusion therapy.
10. Estimated glomerular filtration rate less than 90 mL/min/1.73 m2.
11. Active liver disease or hepatic dysfunction.
12. History of a medical condition associated with an increased risk of bleeding.
13. History of any major surgery within 6 months.
14. History of alcoholism or drug/chemical abuse within 1 year prior to check-in.
15. Use of tobacco- or nicotine-containing products within 6 months prior to check-in.
16. Positive test for illicit drugs and/or tetrahydrocannabinol/cannabinoids at check-in.
17. Female participants with a positive serum pregnancy test.
18. Female participants who are lactating/breastfeeding.
19. Male participants with partners who are pregnant.
20. Unwilling to adhere to contraceptive requirements.
21. Participant has received a dose of an investigational drug within the past 90 days.
22. Have previously completed or withdrawn from this study or any other study investigating teprotumumab or have previously received the investigational product.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-08-26 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Teprotumumab | Up to Day 85
Area Under the Serum Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Teprotumumab | Up to Day 85
Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf) of Teprotumumab | Up to Day 85

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Up to Day 85
Number of Participants With Serious Adverse Events | Up to Day 85
Number of Participants With Anti-teprotumumab Antibodies | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com